CLINICAL TRIAL: NCT07388732
Title: Effects of Abdominal Massage Applied Once and Twice Daily in Phototherapy-Treated Term Newborns on Bilirubin Levels and Defecation: Randomized Controlled Trial
Brief Title: The Effect of Abdominal Massage on Jaundice and Defecation in Newborn Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/137
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hyper Bilirubinemia; Phototherapy; Jaundice, Neonatal
Keywords: Infant massage; Newborn; Phototherapy; Jaundice; Hyperbilirubinemia; Bilirubin
MeSH Terms: conditions — Jaundice, Neonatal; Jaundice; Hyperbilirubinemia

STUDY DESIGN:
Masking Description: Newborns meeting the sampling criteria were assigned to experimental and control groups using a simple random number table. The study was single-blind because the researchers knew which group the newborns in the sample were in. However, the statistical analysis was double-blind because the statistics for the data were performed by a different person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage-1 Group (Experimental): Babies in Massage-1 received a 10-minute abdominal massage once a day before feeding for three days.
  Interventions: Other: Massage once a day for 3 days.
- Massage-2 Group (Experimental): Babies in the Massage-2 group received a 10-minute abdominal massage twice a day before feeding for three days.
  Interventions: Other: Massage twice a day for 3 days.
- Control Group (No Intervention)

INTERVENTIONS:
Other: Massage once a day for 3 days. — The Vimala Massage Application, before massaging, hands were washed and lubricated. The massage began with a patting motion on the newborn's abdomen, followed by clockwise circular movements and semicircles. The massage was then performed in the shapes of an I, inverted L, and U along the abdomen. Finally, a walking movement was performed with the fingertips from the right to the left side of the abdomen. Each movement was repeated six times.
  Arms: Massage-1 Group
Other: Massage twice a day for 3 days. — The Vimala Massage Application, before massaging, hands were washed and lubricated. The massage began with a patting motion on the newborn's abdomen, followed by clockwise circular movements and semicircles. The massage was then performed in the shapes of an I, inverted L, and U along the abdomen. Finally, a walking movement was performed with the fingertips from the right to the left side of the abdomen. Each movement was repeated six times.
  Arms: Massage-2 Group

SUMMARY:
Hyperbilirubinemia is a common condition in term newborns and is often treated with phototherapy. It is thought that abdominal massage may increase bowel movements, thereby increasing the frequency of defecation and supporting bilirubin excretion.

This randomized controlled trial aimed to evaluate the effect of abdominal massage, applied once or twice daily using the Vimala technique, on transcutaneous bilirubin levels and defecation frequency in hyperbilirubinemia-affected term newborns receiving phototherapy in the neonatal intensive care unit.

The study was conducted in the neonatal intensive care unit of a university hospital between February 29, 2020, and August 17, 2023. A total of 35 newborns meeting the inclusion criteria were randomly divided into three groups. Group Massage-1 received 10 minutes of abdominal massage once daily before feeding for three days (n=12). Group Massage-2 received massage twice daily for the same duration (n=10). The control group received routine care (n=13).

ELIGIBILITY:
Inclusion Criteria:

* Term newborns (37-42 weeks gestation)
* 2-10 days postpartum
* Diagnosed with hyperbilirubinemia
* Receiving phototherapy
* Fully orally fed.

Exclusion Criteria:

* Newborns with ABO incompatibility or Rh incompatibility.
* Diagnosed with direct hyperbilirubinemia.
* Genetic/metabolic diseases
* Infections within 24 hours
* With a need for fluid replacement
* Having skin anomalies
* Having abdominal disorders and surgery.

Ages: 2 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-02-29 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
A transcutaneous bilirubin levels | 6 hours after phototherapy
Defecation | Diapers were changed a total of 8 times a day. Defecation outcome was assessed in 24-hour intervals for 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Kütahya, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No